CLINICAL TRIAL: NCT00067132
Title: Adjuvant Nutrition for Critically Ill Trauma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R43DK061818 (completed); MTI-UNR-001; 1R43DK061818 (NIH)
Record Dates: First submitted 2003-08-11; First posted 2003-08-13 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

INTERVENTIONS:
Procedure: Juven (nutritional), HMB (nutritional)

SUMMARY:
Of the four million trauma cases each year that will require hospitalization, 200,000 will be classified as severe trauma. During the hospital stay, malnutrition is a major complication in about 50% of the patient population. The result is muscle wasting which is a major risk factor for increased morbidity and mortality. In this study we postulate that supplementation with beta-hydroxy-beta-methylbutyrate (HMB), arginine and glutamine (HMB/Arg/Gln)or HMB alone to these severely traumatized patients can stem the loss of muscle tissue and whole body nitrogen and in turn decrease morbidity and mortality. This hypothesis is based on two recent studies showing the same nutritional mixture of HMB/Arg/Gln can reverse the muscle wasting associated with AIDS and Cancer. The hypermetabolic state seen in AIDS and cancer have a similar multifactorial etiology as seen in trauma. There is an increase in the mobilization of fat and muscle, increased or normal metabolic rate, increased protein breakdown, and an increased or normal glucose turnover. In addition, HMB alone has been shown to reduce nitrogen loss, decrease muscle proteolysis and muscle damage within the first 48 hours to three weeks after initiating supplementation during a strenuous exercise program. Male and female patients (n=100) will be recruited at the time of admittance to the Trauma ICU with an ISS of greater than 18. Patients who meet the inclusion/exclusion criteria will be randomized to receive either 1) standard tube feed plus HMB/Arg/Gln, 2) standard tube feed plus HMB alone, or 3)standard tube feed (control) in a double-blinded fashion. Clinical outcomes measures will be assessed through out the hospital stay and on an outpatient basis at weeks 4 and 12. Muscle proteolysis and nitrogen economy will be evaluated on daily basis while in the hospital and after 4 weeks on an out patient basis. If as expected, Phase I results confirm the effectiveness of the nutrient mixture in trauma patients, expanded multicenter studies will be proposed in Phase II.

DETAILED DESCRIPTION:
OBJECTIVES:

To compare the effectiveness of immediate nutritional intervention with either HMB, arginine, and glutamine or HMB alone with that of a placebo supplement in critically ill trauma patients on:

* decreasing muscle protein turnover and nitrogen loss
* improving nutritional status,
* improving clinical outcomes,
* preventing total body weight and skeletal muscle loss and
* improving immune status

OUTLINE:

This is a double blind, placebo-controlled randomized clinical study. After receiving informed consent for participation in the study from the next of kin, patients will be randomly assigned to one of the 3 treatment arms:

Arm 1: Standard tube feed plus a nutritional supplement supplying 3 grams of HMB, 14 grams of arginine and 14 grams of glutamine per day. The supplement will be divided into two equal dosages with one dose being given in the morning and one dose given in the evening.

Arm 2: Standard tube feed plus a nutritional supplement supplying 3 grams of HMB. This nutritional supplement will contain gelatin and non-essential amino acids to be isonitrogenous with the supplement in Arm 1. The supplement will also be divided into two equal dosages with one dose being given in the morning and one dose given in the evening.

Arm 3: Standard tube feed plus a nutritional supplement supplying a mixture of gelatin and amino acids to be isonitrogenous with the supplement in Arm 1. The supplement will again be divided into two equal dosages with one dose being given in the morning and one dose given in the evening.

Patients will receive the nutritional supplements for a period of 4 weeks. If a patient leaves the hospital or ICU before that time and/or discontinues the enteral nutrition support, the supplements will be continued orally for the full 4-week period.

Several clinical outcome measures will be followed such as hospital length of stay, ICU length of stay, mortality, number of ventilator days, and incidence of infectious complications. Clinical outcomes will be assessed during the hospital stay and at 4 and 12 weeks. Muscle protein metabolism will be measured during the hospital stay and at 4 weeks. Nutritional status while hospitalized will be assessed by serum pre-albumin levels on days 0,1, 3, 7, and 14. White blood count, number of confirmed infections and C-Reactive Protein levels will serve as proxies for immune status.

ELIGIBILITY:
Inclusion Criteria

* Critically injured trauma patients with an Injury Severity Score (ISS) >18
* Candidate for enteral feeding
* Life expectancy >48 hours
* Total Bilirubin less than or equal to 2.5 mg/dl
* Serum Creatinine less than 3.0 mg/dl.
* Must be able to start supplements within 72 h
* Patient must reside in geographical area of Las Vegas, Nevada

Exclusion Criteria

* Pregnant
* Genetic or immune disorder
* Known hepatitis
* 3rd degree burns involving more than 15% of the body
* Use of other investigational drugs
* Steroid use
* Malignancy
* HIV
* Congestive heart failure
* Inflammatory bowel disease
* Implanted pacemaker or defibrillator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: John A Rathmacher, Ph.D., Principal Investigator — Metabolic Technologies Inc.
Locations (1):
- University Medical Trauma Center/UNSOM, Las Vegas, Nevada, United States

REFERENCES:
- [Background] May PE, Barber A, D'Olimpio JT, Hourihane A, Abumrad NN. Reversal of cancer-related wasting using oral supplementation with a combination of beta-hydroxy-beta-methylbutyrate, arginine, and glutamine. Am J Surg. 2002 Apr;183(4):471-9. doi: 10.1016/s0002-9610(02)00823-1. PMID 11975938
- [Background] Clark RH, Feleke G, Din M, Yasmin T, Singh G, Khan FA, Rathmacher JA. Nutritional treatment for acquired immunodeficiency virus-associated wasting using beta-hydroxy beta-methylbutyrate, glutamine, and arginine: a randomized, double-blind, placebo-controlled study. JPEN J Parenter Enteral Nutr. 2000 May-Jun;24(3):133-9. doi: 10.1177/0148607100024003133. PMID 10850936
- [Background] Panton LB, Rathmacher JA, Baier S, Nissen S. Nutritional supplementation of the leucine metabolite beta-hydroxy-beta-methylbutyrate (hmb) during resistance training. Nutrition. 2000 Sep;16(9):734-9. doi: 10.1016/s0899-9007(00)00376-2. PMID 10978853
- [Background] Nissen S, Sharp R, Ray M, Rathmacher JA, Rice D, Fuller JC Jr, Connelly AS, Abumrad N. Effect of leucine metabolite beta-hydroxy-beta-methylbutyrate on muscle metabolism during resistance-exercise training. J Appl Physiol (1985). 1996 Nov;81(5):2095-104. doi: 10.1152/jappl.1996.81.5.2095. PMID 8941534
- [Background] Williams JZ, Abumrad N, Barbul A. Effect of a specialized amino acid mixture on human collagen deposition. Ann Surg. 2002 Sep;236(3):369-74; discussion 374-5. doi: 10.1097/00000658-200209000-00013. PMID 12192323